CLINICAL TRIAL: NCT02762994
Title: International Multi-center Comparative Randomized Clinical Trial to Evaluate Efficacy and Safety of Multiple Subcutaneous Injections of BCD-085 in Various Doses in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: International Clinical Trial to Evaluate Efficacy and Safety of Multiple Subcutaneous Injections of BCD-085 in Various Doses in Patients With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BCD-085-2
Record Dates: First submitted 2016-04-01; First posted 2016-05-05 (Estimated); Results first posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-02

CONDITIONS: Psoriasis
Keywords: interleukin 17; monoclonal antibody; psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BCD-085, 40 mg (Experimental): Patient will receive 40 mg of BCD-085 subcutaneously at weeks 0, 1, 2, 4, 6, 8, 10.
  Interventions: Drug: BCD-085
- BCD-085, 80 mg (Experimental): Patient will receive 80 mg of BCD-085 subcutaneously at weeks 0, 1, 2, 4, 6, 8, 10.
  Interventions: Drug: BCD-085
- BCD-085, 120 mg (Experimental): Patient will receive 120 mg of BCD-085 subcutaneously at weeks 0, 1, 2, 4, 6, 8, 10.
  Interventions: Drug: BCD-085
- Placebo (Placebo Comparator): Patient will receive placebo subcutaneously at weeks 0, 1, 2, 4, 6, 8, 10.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BCD-085
  Other Names: monoclonal antibody to interleukin 17
  Arms: BCD-085, 120 mg; BCD-085, 40 mg; BCD-085, 80 mg
Other: Placebo
  Arms: Placebo

SUMMARY:
BCD-085-2 is a next step in clinical investigation of BCD-085. BCD-085 is a monoclonal antibody to interleukin 17. During BCD-085-2 trial patients with moderate to severe plaque psoriasis, in whom poor response to previous treatment including UV-therapy and biologic drugs was registered, will receive 40, 80 or 120 mg of BCD-085 subcutaneously at weeks 0, 1, 2, 4, 6, 8, 10. Efficacy and safety parameters will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age between 18 and 65 years
* Diagnosis of plaque psoriasis with stable course of the disease during last 6 months prior to enrollment in the study.
* Patient have had at least 1 course of phototherapy or systemic therapy of psoriasis or are candidates for such treatment.
* BSA affected by psoriasis ≥ 10%, PASI score ≥ 12, sPGA score ≥ 3.
* If patient have had biologic therapy for at least 3 months, there was no positive results of such treatment or patient revealed intolerance to the drug. This therapy must be discontinued at least 12 weeks before enrollment in the study.
* Female patients have negative urine pregnancy test.
* Patient has no history of tuberculosis.
* Patients have negative results of Diaskintest.
* Patient has no history of alcohol or drug abuse.
* Patients are able to perform all procedures planed by protocol.
* Patients are ready for contraception with reliable methods starting 2 weeks before entering the study, and up to 4 weeks after the last dose of study drug.

Exclusion Criteria:

* Subject diagnosed with erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, medication-induced psoriasis, or other skin conditions at the time of the screening visit (e.g., eczema) that would interfere with evaluations of the effect of investigational product on psoriasis.
* Previous receipt of anti-interleukin 17 drugs or anti-interleukin 17 receptor drugs.
* Prior use of two or more biologics to tumor necrosis factor alfa.
* Prior use of two or more biologics to other targets.
* Previous receipt of monoclonal antibodies if they were cancelled less that in 12 weeks before signing informed consent.
* Patient is taking corticosteroids for up to 4 weeks in a dose more than 10 mg (recalculated to prednisolone) before signing informed consent and during screening, or in a dose less than 10 mg (recalculated to prednisolone) if it was not stable.
* Prior use of disease-modifying drugs including methotrexate, sulfasalazin and cyclosporin for up to 4 weeks before signing informed consent, if their dose was not stable for up to 4 weeks before signing informed consent and during screening Prior use of live or attenuated vaccines for up to 8 weeks before signing informed consent.
* Prior use of phototherapy including selective phototherapy and photochemotherapy for up to 4 weeks before signing informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-06; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ivanov, PhD, Study Chair — JCS BIOCAD
Locations (1):
- BIOCAD, Saint Petersburg, Strelna, Russia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- BCD-085, 40 mg: Patient will receive 40 mg of BCD-085 subcutaneously at weeks 0, 1, 2, 4, 6, 8, 10.
  BCD-085
- BCD-085, 80 mg: Patient will receive 80 mg of BCD-085 subcutaneously at weeks 0, 1, 2, 4, 6, 8, 10.
  BCD-085
- BCD-085, 120 mg: Patient will receive 120 mg of BCD-085 subcutaneously at weeks 0, 1, 2, 4, 6, 8, 10.
  BCD-085
- Placebo: Patient will receive placebo subcutaneously at weeks 0, 1, 2, 4, 6, 8, 10.
  Placebo
Period: Overall Study
Arm/Group | BCD-085, 40 mg | BCD-085, 80 mg | BCD-085, 120 mg | Placebo
Started | 31 | 31 | 30 | 28
Completed | 30 | 30 | 28 | 26
Not Completed | 1 | 1 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Provided information only of the patients included in the efficacy assessment (114 subjects).
Groups:
- Total: Total of all reporting groups
Arm/Group | BCD-085, 40 mg | BCD-085, 80 mg | BCD-085, 120 mg | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 28 | 26 | 114
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 41.50 [32.00 to 50.00] | 35.00 [29.00 to 45.00] | 45.00 [35.00 to 54.00] | 41.50 [32.00 to 48.00] | 40.50 [32.00 to 50.00]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 6 | 11 | 35
  Male | 23 | 19 | 22 | 15 | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 30 | 30 | 28 | 26 | 114
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Body weight [Median (Inter-Quartile Range); unit: kg] | 82.00 [70.00 to 90.00] | 80.50 [65.00 to 96.00] | 87.25 [76.00 to 100.00] | 77.55 [64 to 85] | 82.00 [70.00 to 93.50]
Height [Median (Inter-Quartile Range); unit: cm] | 178.50 [170.00 to 182.00] | 173.00 [166.00 to 178.00] | 177.00 [169.40 to 182.00] | 175.00 [164.00 to 182.00] | 176.00 [168.00 to 182.00]
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 25.81 [23.70 to 29.09] | 26.85 [23.62 to 29.59] | 29.72 [24.15 to 31.94] | 24.95 [22.95 to 30.12] | 26.23 [23.73 to 30.60]
Number of Women With Child Bearing Potential [Number; unit: participants] — Population: Provided information only of the women enrolled in the study (35 subjects).
  participants
    number analyzed (Participants) | 7 | 11 | 6 | 11 | 35
    (all) | 5 | 8 | 4 | 8 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With PASI 75 Response After 12 Weeks of Therapy
Description: The PASI allows evaluating the extent and severity of skin symptoms of psoriasis. Body is divided into 4 areas for scoring (head, arms, trunk, legs); each area is scored by itself and scores are combined for final PASI: 0 (no disease) to 72 (maximal disease). The proportion of patients with PASI 75 was defined as patients achieving 75% or more improvement at Week 12 of therapy with BCD-085 from baseline.
Time Frame: 12 weeks
Population: The efficacy analysis was planned to include all patients who received at least one dose of BCD-085/placebo and who attended at least one post-dose visit. The efficacy population comprised of 114 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-085, 40 mg | BCD-085, 80 mg | BCD-085, 120 mg | Placebo
Number analyzed (Participants) | 30 | 30 | 28 | 26
Participants | 24 | 25 | 26 | 6

2. Secondary Outcome: Number of Patients With PASI75 Response After 4 and 8 Weeks of Therapy
Description: The PASI allows evaluating the extent and severity of skin symptoms of psoriasis. Body is divided into 4 areas for scoring (head, arms, trunk, legs); each area is scored by itself and scores are combined for final PASI: 0 (no disease) to 72 (maximal disease). The proportion of patients with PASI 75 was defined as patients achieving 75% or more improvement from baseline.
Time Frame: Week 4, Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- BCD-085, 40 mg: Patients will receive 40 mg of BCD-085 subcutaneously at weeks 0, 1, 2, 4, 6, 8, 10.
  BCD-085
- BCD-085, 80 mg: Patients will receive 80 mg of BCD-085 subcutaneously at weeks 0, 1, 2, 4, 6, 8, 10.
  BCD-085
- BCD-085, 120 mg: Patients will receive 120 mg of BCD-085 subcutaneously at weeks 0, 1, 2, 4, 6, 8, 10.
  BCD-085
- Placebo: Patients will receive placebo subcutaneously at weeks 0, 1, 2, 4, 6, 8, 10.
  Placebo
Arm/Group | BCD-085, 40 mg | BCD-085, 80 mg | BCD-085, 120 mg | Placebo
Number analyzed (Participants) | 30 | 30 | 28 | 26
Participants
  Week 4 | 9 | 10 | 9 | 2
  Week 8 | 22 | 19 | 20 | 3

3. Secondary Outcome: Number of Patients With PASI50 and PASI90 Response After 4, 8 and 12 Weeks of Therapy
Description: The PASI allows evaluating the extent and severity of skin symptoms of psoriasis. Body is divided into 4 areas for scoring (head, arms, trunk, legs); each area is scored by itself and scores are combined for final PASI: 0 (no disease) to 72 (maximal disease). The proportion of patients with PASI 50 and PASI 90 was defined as patients achieving 50% or more and 90% or more improvement from baseline, respectively.
Time Frame: Week 4, Week 8, Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-085, 40 mg | BCD-085, 80 mg | BCD-085, 120 mg | Placebo
Number analyzed (Participants) | 30 | 30 | 28 | 26
Participants
  Proportion of PASI 50 achievers, Week 4 | 19 | 22 | 16 | 4
  Proportion of PASI 50 achievers,Week 8 | 29 | 27 | 27 | 6
  Proportion of PASI 50 achievers,Week 12 | 29 | 30 | 28 | 12
  Proportion of PASI 90 achievers, Week 4 | 1 | 2 | 6 | 0
  Proportion of PASI 90 achievers, Week 8 | 14 | 12 | 15 | 2
  Proportion of PASI 90 achievers, Week 12 | 20 | 18 | 22 | 5

4. Secondary Outcome: Relative Change in PASI Score After 4, 8 and 12 Weeks of Therapy With BCD-085
Description: The PASI allows evaluating the extent and severity of skin symptoms of psoriasis. Body is divided into 4 areas for scoring (head, arms, trunk, legs); each area is scored by itself and scores are combined for final PASI: 0 (no disease) to 72 (maximal disease).
  Relative (percentage) change in PASI score from baseline (screening) is calculated as 100 x (baseline value - time point t value) / (baseline value)
Time Frame: Week 4, Week 8, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | BCD-085, 40 mg | BCD-085, 80 mg | BCD-085, 120 mg | Placebo
Number analyzed (Participants) | 30 | 30 | 28 | 26
percent change
  Mean percentage change from baseline in PASI score at Week 4 | 61.309 (23.423) | 58.855 (27.382) | 59.524 (26.251) | 26.277 (25.933)
  Mean percentage change from baseline in PASI score at Week 8 | 82.148 (17.751) | 78.883 (20.350) | 85.012 (16.389) | 36.512 (29.541)
  Mean percentage change from baseline in PASI score at Week 12 | 88.698 (15.670) | 88.682 (13.607) | 92.771 (11.426) | 45.495 (36.892)

5. Secondary Outcome: Relative Change in BSA After 4, 8 and 12 Weeks of Therapy With BCD-085
Description: The area of skin affected by psoriasis (BSA) is estimated with the palm rule. The area of the human palm without fingers corresponds to about 1% of the body surface.
  Relative (percentage) from baseline is calculated as "100 x (baseline value - time point t value) / (baseline value)". If the value decreases from baseline it means improvement.
Time Frame: Week 4, Week 8, Week 12
Population: The efficacy population comprised of 114 patients.
Measure: Mean (Standard Deviation); unit: percentage of BSA
Arm/Group | BCD-085, 40 mg | BCD-085, 80 mg | BCD-085, 120 mg | Placebo
Number analyzed (Participants) | 30 | 30 | 28 | 26
percentage of BSA
  Mean percentage change from baseline in BSA at Week 4 | 43.046 (31.699) | 45.610 (30.987) | 39.948 (35.084) | 13.692 (22.333)
  Mean percentage change from baseline in BSA at Week 8 | 70.479 (29.547) | 67.233 (30.765) | 68.516 (33.657) | 24.075 (32.046)
  Mean percentage change from baseline in BSA at Week 12 | 82.888 (24.699) | 82.811 (19.751) | 82.074 (29.460) | 36.912 (39.447)

6. Secondary Outcome: Relative Change in NAPSI Score After 12 Weeks of Therapy With BCD-085
Description: The NAPSI is used to assign a score to each nail involved, which can vary from 0 to 8. In this study, nail involvement will be assessed only for hands, so the total index of all nails can be from 0 to 80 (only hands). A negative change from baseline indicates improvement.
  Relative (percentage) change in NAPSI score from baseline (screening) is calculated as 100 x (baseline value - time point t value) / (baseline value)
Time Frame: Week 12
Population: This analysis did not include patients who had no nail psoriasis at baseline and who had no worsening of nail psoriasis during the study (patients who had NAPSI = 0 at baseline and at Week 12). The final population for NAPSI assessment comprised 66 patients.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | BCD-085, 40 mg | BCD-085, 80 mg | BCD-085, 120 mg | Placebo
Number analyzed (Participants) | 17 | 18 | 19 | 12
percent change | 25.204 (45.347) | 47.095 (29.800) | 66.370 (29.455) | 7.828 (36.243)

7. Secondary Outcome: Mean Change in Severity of Pruritus Assessed by Visual Analog Scale After 1, 4, 8 and 12 Weeks of Treatment With BCD-085
Description: Mean change in severity of pruritus assessed by visual analog scale (from 0 (no itch) to 100 mm (unbearable itch)) after 1, 4, 8 and 12 weeks of treatment with BCD-085
Time Frame: Week 1, Week 4, Week 8, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BCD-085, 40 mg | BCD-085, 80 mg | BCD-085, 120 mg | Placebo
Number analyzed (Participants) | 30 | 30 | 28 | 26
units on a scale
  Changes in the intensity of pruritus, Week 1 | -19.600 (23.562) | -25.367 (29.678) | -26.071 (29.034) | -14.269 (34.582)
  Changes in the intensity of pruritus, Week 4 | -34.767 (24.996) | -33.700 (31.682) | -43.214 (30.927) | -13.269 (32.863)
  Changes in the intensity of pruritus, Week 8 | -38.533 (25.871) | -35.633 (34.927) | -47.304 (33.431) | -15.538 (34.195)
  Changes in the intensity of pruritus, Week 12 | -39.533 (26.432) | -40.700 (30.563) | -48.214 (30.839) | -18.269 (34.898)

8. Secondary Outcome: Number of Patients With sPGA Response After 4, 8, 12 Weeks of Treatment With BCD-085
Description: The sPGA scale is used to assess the psoriatic lesions in a certain patient from 0 (clear) to 5 (very severe). Within each area, the severity is estimated by three criteria (induration, desquamation, and erythema).
Time Frame: Week 4, Week 8, Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-085, 40 mg | BCD-085, 80 mg | BCD-085, 120 mg | Placebo
Number analyzed (Participants) | 30 | 30 | 28 | 26
Participants
  sPGA score 0 or 1, Week 4 | 10 | 11 | 8 | 2
  sPGA score 0 or 1, Week 8 | 21 | 19 | 21 | 4
  sPGA score 0 or 1, Week 12 | 25 | 27 | 25 | 8

9. Secondary Outcome: Mean Change in Quality of Life Assessed by SF-36 After 4, 8 and 12 Weeks of Treatment With BCD-085
Description: SF-36 is a standardized participant-administered measure designed to evaluate 8 domains of functional health and well being with 2 components (physical health score [PH] and mental component score [MH]). Both scores range from 0 to 100, with higher scores indicating better levels of function and/or better health.
Time Frame: Week 4, Week 8, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BCD-085, 40 mg | BCD-085, 80 mg | BCD-085, 120 mg | Placebo
Number analyzed (Participants) | 30 | 30 | 28 | 26
units on a scale
  Changes of the PH score from baseline, Week 4 | 3.740 (8.929) | 1.957 (8.691) | 6.943 (9.347) | 2.923 (8.185)
  Changes of the PH score from baseline, Week 8 | 4.763 (9.311) | 3.647 (8.886) | 7.457 (9.115) | 0.992 (10.703)
  Changes of the PH score from baseline, Week 12 | 5.117 (8.731) | 1.820 (10.255) | 7.804 (8.574) | 3.465 (9.437)
  Changes of the MH score from baseline, Week 4 | 6.633 (7.020) | 7.387 (9.915) | 4.196 (11.329) | 3.327 (12.181)
  Changes of the MH score from baseline, Week 8 | 8.773 (9.176) | 8.443 (10.287) | 6.364 (9.946) | 2.792 (9.677)
  Changes of the MH score from baseline, Week 12 | 10.437 (8.939) | 8.693 (10.551) | 5.686 (9.925) | 3.004 (11.361)

10. Secondary Outcome: Mean Change in Quality of Life Assessed by DLQI After 4, 8 and 12 Weeks of Treatment With BCD-085
Description: The Dermatology Life Quality Index (DLQI) is a 10-item self-reported survey, which addresses feelings, daily activities, leisure, work, school, personal relationships, and treatment. Each question was assessed using a 3-point scale, where score 3 means "very much", score 2 means "a lot", score 1 - "a little", and score 0 - "not at all". If more than two questions were left unanswered, the questionnaire was considered invalid. A total score was calculated by summing the score of all items (total maximum score is 30; total minimum score is 0). The higher score representing greater health-related quality of life impairment.
  The mean score change was estimated as the difference between the DLQI at baseline and at the assessed visit (the baseline score was subtracted from the visit score).
Time Frame: Week 4, Week 8, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BCD-085, 40 mg | BCD-085, 80 mg | BCD-085, 120 mg | Placebo
Number analyzed (Participants) | 30 | 30 | 28 | 26
units on a scale
  Changes of the DLQI score, Week 4 | -9.833 (7.292) | -9.000 (6.988) | -8.143 (5.662) | -4.308 (7.121)
  Changes of the DLQI score, Week 8 | -11.967 (7.462) | -11.133 (7.380) | -10.679 (5.157) | -4.846 (7.619)
  Changes of the DLQI score, Week 12 | -13.700 (7.901) | -12.333 (7.369) | -10.107 (7.809) | -5.654 (7.402)

11. Secondary Outcome: Frequency of AE/SAE
Description: Number of participants with AEs and SAEs was presented. The analysis was performed on safety Population which comprised of all participants who received at least one dose of study treatment.
Time Frame: 14 weeks
Population: The safety analysis included all patients who received at least one dose of BCD-085 (31 in Arm 1, 30 in Arm 2, and 28 in each of arms 3 and 4, with the total number n=117).
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-085, 40 mg | BCD-085, 80 mg | BCD-085, 120 mg | Placebo
Number analyzed (Participants) | 31 | 30 | 28 | 28
Participants
  Any AEs/SAEs | 14 | 11 | 7 | 11
  Therapy-related AEs/SAEs | 6 | 3 | 2 | 3
  AEs, grade 3 | 1 | 1 | 1 | 2
  Therapy-related AEs, grade 3 | 1 | 1 | 0 | 0

12. Secondary Outcome: Frequency of Local Reactions
Description: Number of participants with local reactions was presented. The analysis was performed on safety Population which comprised of all participants who received at least one dose of study treatment.
Time Frame: 14 weeks
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-085, 40 mg | BCD-085, 80 mg | BCD-085, 120 mg | Placebo
Number analyzed (Participants) | 31 | 30 | 28 | 28
Participants | 1 | 0 | 0 | 0

13. Secondary Outcome: Frequency of AE/SAE Grade 4 CTCAE 4.03
Description: Number of participants with AEs/SAEs grade 4 CTCAE 4.03 was presented. The analysis was performed on safety Population which comprised of all participants who received at least one dose of study treatment.
Time Frame: 14 weeks
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-085, 40 mg | BCD-085, 80 mg | BCD-085, 120 mg | Placebo
Number analyzed (Participants) | 31 | 30 | 28 | 28
Participants
  Any AEs, grade 4 | 0 | 0 | 0 | 0
  Any SAEs | 0 | 0 | 0 | 0

14. Secondary Outcome: Frequency of Withdrawal Due to AE/SAE
Description: Number of participants who withdrew due to AEs/SAEs was presented. The analysis was performed on safety Population which comprised of all participants who received at least one dose of study treatment.
Time Frame: 14 weeks
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-085, 40 mg | BCD-085, 80 mg | BCD-085, 120 mg | Placebo
Number analyzed (Participants) | 31 | 30 | 28 | 28
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 month
Description: The safety analysis included the data from all patients received at least one dose of BCD-085/placebo. 3 patients were removed from the safety analysis because they recalled their informed consent before the first dose.
  Aggravation, worsening, and symptoms of the plaque psoriasis were not reportable as AEs. If hospitalization was due to aggravation or worsening of psoriasis it was not reportable as an SAE.
Arm/Group | BCD-085, 40 mg | BCD-085, 80 mg | BCD-085, 120 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30 | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 14/31 | 11/30 | 7/28 | 11/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCD-085, 40 mg (N=31) | BCD-085, 80 mg (N=30) | BCD-085, 120 mg (N=28) | Placebo (N=28)
ARVI (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Conjuctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ESR increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lymphocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Total bilirubin increased (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
GGT increased (Hepatobiliary disorders) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
AST increased (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
ALT increased (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Arterial BP increased (Vascular disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Systolic BP increased (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LDH increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flu-like symptoms (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/94/NCT02762994/SAP_000.pdf
  • Study Protocol (2016-07-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT02762994/Prot_001.pdf